CLINICAL TRIAL: NCT03228433
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Oral Single Dose Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-418 in Healthy Subjects
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetics of Ascending Oral Single Dose of TAK-418 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-418-1001; U1111-1195-7777 (Registry Identifier: WHO)
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-08

CONDITIONS: Healthy Participants
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-418

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: TAK-418 5 mg (Experimental): TAK-418 5 milligram (mg), capsule, orally, once on Day 1.
  Interventions: Drug: TAK-418
- Cohort 2: TAK-418 15 mg (Experimental): TAK-418 15 mg, capsule, orally, once on Day 1. Actual dose of TAK-418 may vary based on safety, tolerability and PK data from previous Cohorts.
  Interventions: Drug: TAK-418
- Cohort 3: TAK-418 30 mg Fasted + TAK-418 30 mg Fed (Experimental): TAK-418 30 mg, capsule, in fasted state, orally, once on Day 1, followed by a 28-day washout period, further followed by TAK-418 30 mg, capsule, in fed state, orally, once on Day 1. Actual dose of TAK-418 may vary based on safety, tolerability and PK data from previous Cohorts.
  Interventions: Drug: TAK-418
- Cohort 4: TAK-418 40 mg (Experimental): TAK-418 40 mg, capsule, orally, once on Day 1. Actual dose of TAK-418 may vary based on safety, tolerability and PK data from previous Cohorts.
  Interventions: Drug: TAK-418
- Cohort 5: TAK-418 60 mg (Experimental): TAK-418 60 mg, capsule, orally, once on Day 1. Actual dose of TAK-418 may vary based on safety, tolerability and PK data from previous Cohorts.
  Interventions: Drug: TAK-418
- Cohorts 1-5: Placebo (Placebo Comparator): TAK-418 placebo-matching, capsule, orally, once on Day 1.
  Interventions: Drug: TAK-418 Placebo

INTERVENTIONS:
Drug: TAK-418 — TAK-418 Capsule.
  Arms: Cohort 1: TAK-418 5 mg; Cohort 2: TAK-418 15 mg; Cohort 3: TAK-418 30 mg Fasted + TAK-418 30 mg Fed; Cohort 4: TAK-418 40 mg; Cohort 5: TAK-418 60 mg
Drug: TAK-418 Placebo — TAK-418 placebo-matching capsules.
  Arms: Cohorts 1-5: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of TAK-418 following single oral doses in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-418. TAK-418 is being tested in healthy participants in order to evaluate the safety, tolerability, and pharmacokinetics (PK) of single oral doses.

The study will enroll approximately 40 healthy participants. The study consists of equally divided 5 sequential cohorts of 8 participants each. In each of the following cohorts, 6 participants will be randomized to receive TAK-418 and 2 participants will receive matching placebo-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Cohort 1: TAK-418 5 mg
* Cohort 2: TAK-418 15 mg
* Cohort 3: TAK-418 30 mg Fasted + TAK-418 30 mg Fed
* Cohort 4: TAK-418 40 mg
* Cohort 5: TAK-418 60 mg

All participants will be asked to take TAK-418 or placebo-matching capsule once on Day 1 in each cohort. A washout period of 28-days will be maintained between the doses in Cohort 3.

This single center trial will be conducted in the United States. Participants in this study will be assigned to one of 5 possible dose cohorts. Male participants will return for additional outpatient visits on Days 91 and 93 (+/- 7 days) and may return for outpatient visits on Days 182 and 184 (+/- 7 days) (depending on results from the Day 93 Visit).

ELIGIBILITY:
Inclusion Criteria:

1. Is a male or female participants with a body mass index (BMI) within the range of 18.5 -30.0 kilogram per square meter (kg/m^2) at the Screening Visit.
2. Is a nonsmoker who has not used tobacco or nicotine-containing products (example, nicotine patch) for at least 6 months before trial drug administration of the initial dose of trial drug or invasive procedure.
3. Must be judged to be in good health by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead ECG, and vital sign measurements performed at the Screening Visit and before administration of the initial dose of trial drug or invasive procedure as per principal investigator's judgment.
4. Female subjects with no childbearing potential, defined by at least 1 of the following criteria:

   * Postmenopausal (defined as 12 months of spontaneous amenorrhea in women aged greater than [>]45 years, 6 months of spontaneous amenorrhea in women aged >45 years with serum follicle-stimulating hormone [FSH] levels >40 milli-international units per milliliter [mIU/mL]). Appropriate documentation of FSH levels is required.
   * Surgically sterile by hysterectomy and/or bilateral oophorectomy with appropriate documentation of surgical procedure.
   * Had a tubal ligation with appropriate documentation of surgical procedure.
   * Has a congenital condition resulting in no uterus.

Exclusion Criteria:

1. Has had major surgery, donated or lost 1 unit of blood (approximately 500 milliliter [mL]) within 4 weeks before the Screening Visit.
2. Has a risk of suicide according to the investigator's clinical judgment per the Columbia-Suicide Severity Rating Scale at Screening or has made a suicide attempt in the 6 months before Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2018-05-12 (Actual); Study Completion 2018-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- PAREXEL International, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Yin W, Arkilo D, Khudyakov P, Hazel J, Gupta S, Quinton MS, Lin J, Hartman DS, Bednar MM, Rosen L, Wendland JR. Safety, pharmacokinetics and pharmacodynamics of TAK-418, a novel inhibitor of the epigenetic modulator lysine-specific demethylase 1A. Br J Clin Pharmacol. 2021 Dec;87(12):4756-4768. doi: 10.1111/bcp.14912. Epub 2021 Jun 10. PMID 33990969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at single site in the United States from 21 July 2017 to 12 May 2018.
Pre-assignment Details: Healthy participants were randomized to receive TAK-418 or matching placebo in Cohorts 1 to 5.
Groups:
- Cohort 2: TAK-418 15 mg: TAK-418 15 mg, capsule, orally, once on Day 1.
- Cohort 3: TAK-418 30 mg Fasted + TAK-418 30 mg Fed: TAK-418 30 mg, capsule, in fasted state, orally, once on Day 1, followed by a 28-day washout period, further followed by TAK-418 30 mg, capsule, in fed state, orally, once on Day 1.
- Cohort 4: TAK-418 40 mg: TAK-418 40 mg, capsule, orally, once on Day 1.
- Cohort 5: TAK-418 60 mg: TAK-418 60 mg, capsule, orally, once on Day 1.
Period: Overall Study
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3: TAK-418 30 mg Fasted + TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Started | 10 | 6 | 6 | 6 | 6 | 6
Completed | 9 | 6 | 6 | 5 | 6 | 6
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Positive alcohol test | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Cohort 1: TAK-418 5 mg: TAK-418 5 mg, capsule, orally, once on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3: TAK-418 30 mg Fasted + TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (9.63) | 37.2 (10.42) | 33.3 (10.80) | 40.0 (10.60) | 33.2 (6.49) | 38.7 (10.03) | 36.5 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 1 | 0 | 3 | 8
  Male | 8 | 4 | 6 | 5 | 6 | 3 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 0 | 1 | 1 | 7
  Not Hispanic or Latino | 9 | 4 | 4 | 6 | 5 | 5 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 2 | 1 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 5 | 1 | 1 | 0 | 2 | 0 | 9
  White | 4 | 4 | 3 | 4 | 2 | 5 | 22
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 6 | 6 | 6 | 6 | 40
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 81.2 (12.34) | 76.0 (13.58) | 81.8 (6.83) | 82.5 (4.22) | 80.0 (12.43) | 76.1 (15.23) | 79.8 (11.0)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 173.4 (8.66) | 171.0 (8.10) | 174.8 (3.19) | 172.5 (5.09) | 181.2 (5.08) | 171.5 (11.78) | 174.0 (7.89)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.94 (3.065) | 25.82 (2.440) | 26.83 (2.835) | 27.83 (2.414) | 24.32 (2.988) | 25.73 (2.992) | 26.32 (2.864)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline Up to Day 184
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Cohort 3A: TAK-418 30 mg Fasted: TAK-418 30 mg, capsule, in fasted state, orally, once on Day 1.
- Cohort 3B: TAK-418 30 mg Fed: TAK-418 30 mg, capsule, in fed state, orally, once on Day 1.
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 5 | 6 | 6
participants | 4 | 2 | 2 | 3 | 1 | 3 | 3

2. Primary Outcome: Number of Participants Who Discontinued Due to an Adverse Event (AE)
Time Frame: Baseline Up to Day 184
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 5 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Meet the Markedly Abnormal Criteria for Neurological Assessment Measurements at Least Once Post Dose
Time Frame: Baseline Up to Day 184
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 5 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Time Frame: Baseline Up to Day 184
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 5 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose
Time Frame: Baseline Up to day 184
Population: The safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 5 | 6 | 6
participants
  Diastolic blood pressure less than (<) 50 mmHg | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Systolic blood pressure < 85 mmHg | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Temperature < 35.6 degrees celsius (°C) | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Temperature greater than (>) 37.7 (°C) | 0 | 0 | 0 | 0 | 0 | 0 | 2

6. Primary Outcome: Number of Participants Who Meet the Markedly Abnormal Criteria for Safety 12-lead Electrocardiogram (ECG) Parameters at Least Once Post Dose
Time Frame: Baseline Up to Day 14
Measure: Number; unit: participants
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 5 | 6 | 6
participants
  ECG ventricular rate(Beats/ minute) | 1 | 2 | 1 | 0 | 0 | 0 | 0
  QT interval (Milliseconds) | 0 | 1 | 0 | 0 | 0 | 0 | 1

7. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration of TAK-418F (TAK-418 Free Base)
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The pharmacokinetic analysis set included all participants who received at least 1 dose of study drug and had at least one measurable plasma concentration or amount of drug in urine for TAK-418-F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
hour nanogram per milliliter (h*ng/mL) | 77.3 (47.1) | 290.4 (21.8) | 649.4 (8.5) | 616.2 (23.1) | 674.1 (27.0) | 1576.3 (33.5)
Statistical Analysis 1: Comparison: Cohort 3A: TAK-418 30 mg Fasted vs Cohort 3B: TAK-418 30 mg Fed; Test type: Equivalence — A linear mixed effect model on the natural log-transformed parameters was performed with a fixed effect for regimen and random effect for participant. The least squares(LS) means and difference of least squares (LS) means for the log-transformed parameters were exponentiated to obtain the point estimates (Geometric LS means) of the food effect and 90% confidence intervals (CIs); Least Squares (LS) Mean Difference = 0.951, 90% CI 2-sided [0.823 to 1.099]
Statistical Analysis 2: Comparison: Cohort 1: TAK-418 5 mg vs Cohort 2: TAK-418 15 mg vs Cohort 3A: TAK-418 30 mg Fasted vs Cohort 4: TAK-418 40 mg vs Cohort 5: TAK-418 60 mg; Test type: Equivalence — A linear regression model (power model), log (ln) (parameter) equal to (=) intercept plus (+) slope*ln (dose), was fit to describe the relationship between each parameter and the corresponding dose levels. Dose Proportionality was declared if the 90% CI of the slope lied entirely within the critical region as defined by 1 - ln(0.8) per (/)l n(r) to 1 + ln(1.25)/ln(r), where r was the ratio of the highest and lowest dose in the study; Slope = 1.14, 90% CI 2-sided [1.04 to 1.25]

8. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-418F
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
h*ng/mL | 84.9 (47.4) | 296.3 (22.1) | 659.6 (8.0) | 626.0 (22.7) | 681.0 (26.9) | 1519.9 (33.3)
Statistical Analysis 1: Comparison: Cohort 3A: TAK-418 30 mg Fasted vs Cohort 3B: TAK-418 30 mg Fed; Test type: Equivalence — Bioequivalence interval of 627.51 to 659.59; LS Mean Difference = 0.951, 90% CI 2-sided [0.825 to 1.097]
Statistical Analysis 2: Comparison: Cohort 1: TAK-418 5 mg vs Cohort 2: TAK-418 15 mg vs Cohort 3A: TAK-418 30 mg Fasted vs Cohort 4: TAK-418 40 mg vs Cohort 5: TAK-418 60 mg; Test type: Equivalence — A linear regression model (power model), ln (parameter) = intercept + slope*ln (dose), was fit to describe the relationship between each parameter and the corresponding dose levels. Dose Proportionality was declared if the 90% CI of the slope lied entirely within the critical region as defined by 1 - ln (0.8)/l n(r) to 1 + ln (1.25)/ln(r), where r was the ratio of the highest and lowest dose in the study; Slope = 1.11, 90% CI 2-sided [1.00 to 1.22]

9. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-418F
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
nanogram per millilitre (ng/mL) | 21.54 (35.9) | 61.90 (26.6) | 163.64 (20.9) | 94.93 (33.8) | 155.32 (34.3) | 321.52 (14.1)
Statistical Analysis 1: Comparison: Cohort 3A: TAK-418 30 mg Fasted vs Cohort 3B: TAK-418 30 mg Fed; Test type: Equivalence — A linear mixed effect model on the natural log-transformed parameters was performed with a fixed effect for regimen and random effect for participant. The LS means and difference of LS means for the log-transformed parameters were exponentiated to obtain the point estimates (Geometric LS means) of the food effect and 90% confidence intervals CIs; LS Mean Difference = 0.580, 90% CI 2-sided [0.431 to 0.781]
Statistical Analysis 2: Comparison: Cohort 1: TAK-418 5 mg vs Cohort 2: TAK-418 15 mg vs Cohort 3A: TAK-418 30 mg Fasted vs Cohort 4: TAK-418 40 mg vs Cohort 5: TAK-418 60 mg; Test type: Equivalence — [test comment as in outcome 8, analysis 2]; Slope = 1.06, 90% CI [0.96 to 1.17]

10. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-418F
Description: The pharmacokinetic analysis set included all participants who received at least 1 dose of study drug and had at least one measurable plasma concentration or amount of drug in urine for TAK-418-F.
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6
hour | 1.000 [0.98 to 1.02] | 1.000 [1.00 to 2.00] | 1.000 [0.50 to 1.00] | 3.000 [1.50 to 3.02] | 1.250 [1.00 to 1.52] | 1.000 [1.00 to 1.00]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of the study drug up to Day 184
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohorts 1-5: Placebo | Cohort 1: TAK-418 5 mg | Cohort 2: TAK-418 15 mg | Cohort 3A: TAK-418 30 mg Fasted | Cohort 3B: TAK-418 30 mg Fed | Cohort 4: TAK-418 40 mg | Cohort 5: TAK-418 60 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/10 | 2/6 | 2/6 | 3/6 | 1/5 | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1-5: Placebo (N=10) | Cohort 1: TAK-418 5 mg (N=6) | Cohort 2: TAK-418 15 mg (N=6) | Cohort 3A: TAK-418 30 mg Fasted (N=6) | Cohort 3B: TAK-418 30 mg Fed (N=5) | Cohort 4: TAK-418 40 mg (N=6) | Cohort 5: TAK-418 60 mg (N=6)
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion .

DOCUMENTS (2):
  • Study Protocol (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03228433/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03228433/SAP_001.pdf